CLINICAL TRIAL: NCT01363921
Title: Effect of High Cut-off Membranes on Cardiovascular Function in Patients With End-stage Renal Disease (HICOCARD)
Brief Title: Effect of HCO1100 on Cardiovascular Function
Acronym: HicoCARD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient patient recruiting
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HicoCARD 1481
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Disease; Chronic Kidney Failure
Keywords: CKD5; dialysis; high porous membranes; micro-inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dialysis treatment with HCO1100 (Experimental)
  Interventions: Device: HCO 1100

INTERVENTIONS:
Device: HCO 1100 — Dialysis treatment with HCO1100
  Other Names: High cut-off membrane

SUMMARY:
The purpose of this study is to determine whether high porous membranes are effective in the treatment of cardiovascular events in chronic dialysis patients.

DETAILED DESCRIPTION:
Cardiovascular events are the leading cause of the increased mortality rate of chronic dialysis patients. It is believed that increased micro-inflammation plays an important role in the pathophysiological process of cardiovascular disease. High porous dialysis membranes can better eliminate inflammatory mediators as compared to standard dialysis membranes. In this study, the high porous dialysis membrane HCO1100 is investigated for its potential capability to improve the cardiovascular status of chronic dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Dialysis dependent chronic renal failure (CKD 5) in a stable condition
* Serum albumin at randomisation equal to or above the median of the normal range (pre- dialysis value)

Exclusion Criteria:

* Diabetes mellitus as the disease underlined end stage renal failure
* Haemodynamic instability that precludes unsupported dialysis
* planned surgical interventions <= 4 months at time of inclusion
* known allergy against dialysis membranes
* Significant cardiac disease (atrial fibrillation, myocardial infarction within 6 months; unstable angina pectoris; LV-EF < 30%, clinically significant pericardial disease; cardiac amyloidosis)
* pulmonary disease with chronic hypoxia
* Advanced disease or significant co-morbidity with poor short term prognosis, necessitating palliation and not subject to active or disease specific treatment
* Clinically significant liver dysfunction (bilirubin > 1.8mg/dl (30µmol/L))
* Prior fistula surgery on both arms or other operations or paralysis on both arms
* Known HIV, HCV infection
* Alcoholism
* Active uncontrolled infection
* Pregnancy or lactation
* Inability to give informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes in hyperoxic chemoreflex sensitivity (CHRS) and flow mediated endothelial vasodilatation (FMD) | max 15 weeks
  Changes of CHRS (ms/mmHg) and FMD (%) between pre- and post- treatment phase with study product HCO1100 dialyzer and at 6 weeks follow up after termination of HCO1100 dialyzer treatment phase will be assessed.

SECONDARY OUTCOMES:
Weekly assessment of albumin plasma levels (g/l) | max 15 weeks
  Weekly evaluation of albumin plasma levels (g/l) during the study. Patients with albumin plasma levels below 35g/l will terminate study product (HCO1100 dialyzer) treatment phase and switch to study phase with control standard dialyzer treatment and will be further monitored for 6 weeks. Number of patients with decreased albumin levels below 35g/l , Number of patients with requirement for albumin substitution and absolute albumin drop (g/l) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Floege, MD, Principal Investigator — Med.Klinik II, Universitätsklinikum Aachen
Locations (1):
- Med. Klinik II, Nephrologie und med. Immunologie, Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia, Germany